CLINICAL TRIAL: NCT01645735
Title: A Multicenter, Multinational, Randomized, Double-blind Study to Evaluate the Efficacy and Safety of Ceftaroline Fosamil Versus Ceftriaxone Plus Vancomycin in Adult Subjects With Community-acquired Bacterial Pneumonia at Risk for Infection Due to Methicillin-resistant Staphylococcus Aureus
Brief Title: Evaluation of Ceftaroline Fosamil Versus a Comparator in Adult Subjects With Community-acquired Bacterial Pneumonia (CABP) With Risk for Methicillin-resistant Staphylococcus Aureus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P903-25
Record Dates: First submitted 2012-07-09; First posted 2012-07-20 (Estimated); Results first posted 2016-02-01 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2015-12

CONDITIONS: Infections
Keywords: Infections; Teflaro; cephalosporin; Ceftaroline; antibiotics; pneumonia
MeSH Terms: conditions — Infections; Pneumonia | interventions — Ceftaroline; Ceftriaxone; Vancomycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ceftaroline (Experimental): Ceftaroline fosamil 600 mg Intravenous (IV) administration over 60 minutes, every 8 hours (q8h); dosing to be adjusted for renal function; treatment duration 5 to 14 days
  Interventions: Drug: Ceftaroline fosamil
- Ceftriaxone plus vancomycin (Active Comparator): Ceftriaxone 2 g IV over 30 minutes once per day (q24h) plus vancomycin 15 mg/kg IV every 12 hours (q12h) initially and then dose adjusted based on trough concentrations; treatment duration 5 to 14 days
  Interventions: Drug: Ceftriaxone plus vancomycin

INTERVENTIONS:
Drug: Ceftaroline fosamil — Ceftaroline fosamil 600 mg IV over 60 minutes q8h; treatment duration 5 to 14 days
  Other Names: Teflaro; PPI-0903; TAK-599; TAK599; PPI0903 Teflaro
  Arms: Ceftaroline
Drug: Ceftriaxone plus vancomycin — Ceftriaxone 2g IV over 30 minutes q24h plus vancomycin 15 mg/kg IV q12h initially and then dose adjusted based on trough concentrations; treatment duration 5 to 14 days
  Arms: Ceftriaxone plus vancomycin

SUMMARY:
The purpose of this study is to determine whether ceftaroline is effective and safe for the treatment of patients with Community-acquired Bacterial Pneumonia (CABP) at risk for infection due to Methicillin-resistant Staphylococcus aureus (MRSA).

DETAILED DESCRIPTION:
A Multicenter, Multinational, Randomized, Double-blind Study to Evaluate the Efficacy and safety of Ceftaroline fosamil Versus Ceftriaxone Plus Vancomycin in Adult Subjects with Community-acquired Bacterial Pneumonia at Risk for Infection Due to Methicillin-resistant Staphylococcus aureus.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are required to meet All of the following inclusion criteria:

  1. Male or female, ≥ 18 years old
  2. Presence of CABP requiring hospitalization
  3. Presence of CABP meeting the following criteria:

I. confirmed pneumonia (new or progressive pulmonary) II. Acute illness (≤ 7 days' duration) with at least 3 clinical signs or symptoms consistent with a lower respiratory tract infection

MRSA Risk Factors

• MRSA-positive blood culture or respiratory specimen or a risk factor for MRSA such as a history of colonization with MRSA

Exclusion Criteria:

* Subjects must Not meet any of the following exclusion criteria at baseline:

  1. History of any hypersensitivity or allergic reaction to any β-lactam antimicrobial
  2. Suspected or microbiologically-documented infection with a pathogen known to be resistant to any of the study drugs
  3. Non-infectious causes of pulmonary infiltrates (eg, pulmonary embolism, chemical pneumonitis from aspiration, hypersensitivity pneumonia, congestive heart failure)
  4. More than 24 hours of potentially effective systemic antibacterial therapy for CABP within 96 hours before randomization
  5. End-stage renal disease [Creatinine Clearance (CrCl) < 15], including hemodialysis
  6. Evidence of significant hepatic, hematological, or immunocompromising condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Forest Laboratories Inc, an affiliate of Allergan plc
Locations (31):
- United States (13):
  - Investigational Site, Phoenix, Arizona
  - Investigational Site, Sylmar, California
  - Investigational Site, DeLand, Florida
  - Investigational Site, Chicago, Illinois
  - Investigational Site, Kansas City, Kansas
  - Investigational Site, Royal Oak, Michigan
  - Investigational Site, Minneapolis, Minnesota
  - Investigational Site, St Louis, Missouri
  - Investigational Site, Omaha, Nebraska
  - Investigational Site, Laconia, New Hampshire
  - Investigational Site, Columbus, Ohio
  - Investigational Site, Lima, Ohio
  - Investigational Site, Oklahoma City, Oklahoma
- Investigational Site, Tbilisi, Georgia
- Investigational Site, Mátraháza, Hungary
- Poland (3):
  - Investigational Site, Lodz
  - Investigational Site, Lublin
  - Investigational Site, Wilkowice-Bystra
- Romania (3):
  - Investigational Site, Craiova, Dolj
  - Investigational Site, Bucharest
  - Investigational Site, Iași
- Russia (3):
  - Investigational Site, Moscow
  - Investigational Site, Saint Petersburg
  - Investigational Site, Yaroslavl
- Spain (2):
  - Investigational Site, Alicante
  - Investigational Site, Barcelona
- Ukraine (5):
  - Investigational Site, Dnipropetrovsk
  - Investigational Site, Ivano-Frankivsik
  - Investigational Site, Kharkiv
  - Investigational Site, Kyiv
  - Investigational Site, Zaporizhzhya

REFERENCES:
- See also: Related Info — http://www.cerexa.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Ceftaroline: Ceftaroline fosamil 600 mg IV over 60 minutes q8h; treatment duration 5 to 14 days
- Ceftriaxone Plus Vancomycin: Ceftriaxone 2 g IV q24 plus vancomycin 15 mg/kg IV q12h initially and then dose adjusted based on trough concentrations; treatment duration 5 to 14 days
Period: Overall Study
Arm/Group | Ceftaroline | Ceftriaxone Plus Vancomycin
Started | 32 | 17
Completed | 28 | 16
Not Completed | 4 | 1
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: * Safety: all randomized who received any amount of study drug
  * MITT: all randomized who received any amount of IV study drug & had a confirmed CABP w/risk factors for MRSA (excluding those w/sole atypical pathogen)
  * mMITT: MITT subset, including subjects w/at least 1 typical bacterial pathogen identified from adequate micro specimen at baseline
Groups:
- Ceftaroline: Ceftaroline fosamil 600 mg IV over 60 minutes q8h
- Ceftriaxone Plus Vancomycin: Ceftriaxone 2g IV over 30 minutes q24h plus vancomycin 15 mg/kg IV q12h initially and then dose adjusted based on trough concentrations
- Total: Total of all reporting groups
Arm/Group | Ceftaroline | Ceftriaxone Plus Vancomycin | Total
Number analyzed (Participants) | 32 | 17 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (17.09) | 68.1 (14.14) | 58.3 (17.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 4 | 16
  Male | 20 | 13 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 29 | 17 | 46
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 31 | 17 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Creatinine Clearance [Mean (Standard Deviation); unit: mL/min/1.73 m^2] | 92.47 (52.190) | 66.52 (24.448) | 83.47 (45.978)
PORT Score [Mean (Standard Deviation); unit: units on a scale] — The Pneumonia Outcomes Research Team (PORT) Score is a clinical prediction rule for medical practitioners to calculate the probability of morbidity and mortality among patients with community acquired pneumonia. Based on the patient's age, nursing home resident status, coexisting illnesses, physical examination findings, as well as laboratory and radiographic findings. The PORT score ranges from:
  A low risk of
  Men - Patient's age in years. Women - Patient's age in years minus 10.
  To a high risk of
  Men - Patient's age in years plus 285. Women - Patient's age in years plus 275.
  units on a scale | 89.8 (33.17) | 118.6 (29.47) | 99.8 (34.53)

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response at Study Day 4 in the Modified Intent-to-Treat (MITT) Population
Description: Clinical response was defined as meeting all of the following criteria:
  * Symptom Improvement - Improvement in at least 2 and no worsening of any of the following symptoms compared to baseline:
    * Cough
    * Dyspnea
    * Sputum production
    * Chest pain
  * Clinical Stability (per Infectious Diseases Society of America/American Thoracic Society (IDSA/ATS) guidelines; Mandell et al, 2007):
    * Temperature ≤ 37.8°C
    * Heart rate ≤ 100 beats/min
    * Respiratory rate ≤ 24 breaths/min
    * Systolic blood pressure ≥ 90 mmHg
    * Oxygen saturation ≥ 90%
    * Confusion/disorientation absent
Time Frame: Study Day 4
Population: MITT Population: all randomized subjects who receive any amount of IV study drug and who have a confirmed diagnosis of Community-Acquired Bacterial Pneumonia (CABP) with risk factors for Methicillin-Resistant Staphylococcus aureus (MRSA) (excluding those that have a sole atypical pathogen)
Measure: Number; unit: participants
Groups:
- Ceftriaxone Plus Vancomycin: Ceftriaxone 2 g IV q24 plus vancomycin 15 mg/kg IV q12h initially and then dose adjusted based on trough concentrations
Arm/Group | Ceftaroline | Ceftriaxone Plus Vancomycin
Number analyzed (Participants) | 32 | 17
participants
  Responder | 14 | 8
  Non-Responder | 16 | 8
  Incomplete Data | 2 | 1

2. Primary Outcome: Clinical Outcome at Test of Cure (TOC) in the MITT Population
Description: An assessment of clinical outcome was made by the Investigator at TOC. The clinical outcome categories were:
  Cure: Resolution of all acute signs and symptoms of CABP or improvement to such an extent that no further antimicrobial therapy was required
  Failure: Subjects who meet either of the following criteria:
  * Incomplete resolution or worsening of CABP signs and symptoms or development of new CABP signs or symptoms requiring alternative nonstudy antimicrobial therapy
  * Death in which CABP is contributory
  Indeterminate: Study data are not available for evaluation of efficacy for any reason, including:
  * Death in which CABP is clearly noncontributory
  * Lost to follow-up
  * Extenuating circumstances precluding classification as a cure or failure
  A favorable clinical outcome at Test-of Cure (TOC) was clinical cure.
Time Frame: Test of Cure, an average of 3 weeks
Population: MITT Population: all randomized subjects who receive any amount of IV study drug and who have a confirmed diagnosis of CABP with risk factors for MRSA (excluding those that have a sole atypical pathogen)
Measure: Number; unit: participants
Groups:
- Ceftriaxone Plus Vancomycin: Ceftriaxone 2g IV q24 plus vancomycin 15mg/kg IV q12h initially and then dose adjusted based on trough concentrations
Arm/Group | Ceftaroline | Ceftriaxone Plus Vancomycin
Number analyzed (Participants) | 32 | 17
participants
  Clinical Cure | 27 | 15
  Clinical Failure | 3 | 2
  Indeterminate | 2 | 0

3. Other Pre Specified Outcome: Microbiological Outcomes by Baseline Pathogen at TOC in the Microbiological Modified Intent-to-Treat (mMITT) Population
Description: An overall microbiological outcome was derived based on the subject's baseline pathogen. As no follow-up specimens were collected at the TOC visit for any subjects, all microbiological outcomes were derived based strictly on clinical outcomes, as either presumed eradication (ie, source specimen was not available to culture and the subject was assessed as clinical cure) , presumed persistence (ie, source specimen was not available to culture and the subject was assessed as a clinical failure), or indeterminate (ie, source specimen was not available to culture and the subject's clinical response was assessed as indeterminate).
Time Frame: Test of Cure, an average of 3 weeks
Population: mMITT Population: a subset of the MITT Population, including subjects for whom at least 1 typical bacterial pathogen has been identified from an adequate microbiological specimen at baseline
Measure: Number; unit: participants
Arm/Group | Ceftaroline | Ceftriaxone Plus Vancomycin
Number analyzed (Participants) | 25 | 14
participants
  Presumed eradication | 23 | 12
  Presumed persistence | 0 | 2
  Indeterminate | 2 | 0

4. Other Pre Specified Outcome: Safety Evaluation
Description: Adverse events (AEs), serious adverse events (SAEs), deaths, discontinuation due to AEs
Time Frame: Baseline (Day 0) to Day 49
Population: Safety Population: all randomized subjects who received any amount of IV study drug
Measure: Number; unit: participants
Arm/Group | Ceftaroline | Ceftriaxone Plus Vancomycin
Number analyzed (Participants) | 32 | 17
participants
  Any TEAE | 17 | 9
  Any study drug-related TEAEs | 3 | 2
  Any SAEs | 3 | 2
  Any study drug-related SAEs | 0 | 0
  Discontinuation of IV or oral study drug due to AE | 1 | 1
  Discontinuation of IV study drug only due to AE | 1 | 1
  Deaths | 1 | 0

ADVERSE EVENTS:
Groups:
- Ceftriaxone Plus Vancomycin: Ceftriaxone 2 g IV over 30 minutes q24h plus vancomycin 15 mg/kg IV q12h initially and then dose adjusted based on trough concentrations
Arm/Group | Ceftaroline | Ceftriaxone Plus Vancomycin
Serious Adverse Events (participants affected / at risk) | 3/32 | 2/17
Other Adverse Events (participants affected / at risk) | 9/32 | 9/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ceftaroline (N=32) | Ceftriaxone Plus Vancomycin (N=17)
Angina pectoris (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Computerized tomogram thorax abnormal (Investigations) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ceftaroline (N=32) | Ceftriaxone Plus Vancomycin (N=17)
Anemia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 2
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 1
Edema Peripheral (General disorders) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0
Blood pressure increased (Investigations) | 0 | 1
Body temperature increased (Investigations) | 0 | 1
Neutrophil count increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Headache (Nervous system disorders) | 3 | 1
Disorientation (Psychiatric disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Small number of subjects enrolled

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The data generated in this clinical study are the exclusive property of the Sponsor and are confidential. The Sponsor will make all reasonable efforts to publish the results of the study in an appropriate peer-reviewed journal. Authorship on the primary publication of the results from this study will be based on contributions to study design, enrollment, data analysis, and interpretation of results. Publication of results by the PI will be subject to mutual agreement between the PI and Sponsor.